CLINICAL TRIAL: NCT06361329
Title: A Multicenter, Prospective, Randomized Controlled Clinical Study Comparing the Efficacy of VHAG and Traditional Chemotherapy Regimens in the Treatment of Adult Newly Diagnosed Early Precursor T-cell Acute Lymphoblastic Leukemia (ETP-ALL)
Brief Title: Comparing the Efficacy of VHAG and Traditional Chemotherapy Regimens in Newly Diagnosed ETP-ALL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240030C
Record Dates: First submitted 2024-04-01; First posted 2024-04-11 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-03

CONDITIONS: ETP-ALL
MeSH Terms: interventions — Homoharringtonine; venetoclax; Cytarabine; Granulocyte Colony-Stimulating Factor; Vindesine; Daunorubicin; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VHAG group (Experimental): Venetoclax: 100mg on day 1, 200mg on day 2, and 400mg on days 3-14, if the blast cells in bone marrow were more than 5% on day 14, the patient continued to receive venetoclax 400mg until day 28.
  HHT:1.4 mg/m2,2mg maximum daily, intravenously daily from on d1-7 Cytarabine :10 mg/m2 subcutaneously every 12h on d1-14（d10-d14） G-CSF: 100ug/m2 daily on d1-14 if WBC count <10*10E9/L
  Interventions: Drug: Homoharringtonine; Drug: venetoclax; Drug: Cytarabine; Drug: G-CSF
- Traditional Chemotherapy Regimen group (Active Comparator): * VDCLP regimen
  * VD(/I) CP regimen
  * Hyper CVAD-A regimen
  * VDLP regimen
  Interventions: Drug: Cytarabine; Drug: Vindesine; Drug: Daunorubicin; Drug: cyclophosphamide; Drug: Dexamethasone; Drug: L-ASP

INTERVENTIONS:
Drug: Homoharringtonine — Intravenous infusion
  Arms: VHAG group
Drug: venetoclax — Orally by mouth
  Arms: VHAG group
Drug: Cytarabine — subcutaneous injection or Intravenous infusion
Drug: G-CSF — subcutaneous injection
  Arms: VHAG group
Drug: Vindesine — Intravenous infusion
  Arms: Traditional Chemotherapy Regimen group
Drug: Daunorubicin — Intravenous infusion
  Arms: Traditional Chemotherapy Regimen group
Drug: cyclophosphamide — Intravenous infusion
  Arms: Traditional Chemotherapy Regimen group
Drug: Dexamethasone — Intravenous infusion or orally
  Arms: Traditional Chemotherapy Regimen group
Drug: L-ASP — subcutaneous injection
  Arms: Traditional Chemotherapy Regimen group

SUMMARY:
ETP-ALL is a subtype of T-cell acute lymphoblastic leukemia (T-ALL) with poor outcomes and prognosis. Effective induction therapy is crucial in improving the treatment effect. Based on our laboratory research and clinical practice, the venetoclax plus HAG regimen shows promising efficacy in treating ETP-ALL. Therefore, we plan to conduct a prospective, multicenter Phase III clinical study to evaluate the efficacy of the venetoclax plus HAG regimen in treating newly diagnosed ETP-ALL patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥14 and <75 years old.
* Diagnosed with ETP-ALL (including near-ETP ALL) before enrollment.
* Newly diagnosed patients.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Expected survival of ≥3 months.
* Able to undergo oral treatment with venetoclax.
* No organ dysfunction that would restrict the treatment administered
* Understanding of the study and signing of the informed consent form.
* Men, women of childbearing potential (postmenopausal women must have been amenorrheic for at least 12 months to be considered infertile), and their partners must voluntarily use effective contraception methods as deemed appropriate by the investigator during the treatment period and for at least 12 months after the last dose of the study drug.

Exclusion Criteria:

* Patients who are unable to take venetoclax by mouth;
* Patients with severe heart, lung, liver, kidney, or other organ dysfunction that may restrict their participation in this trial due to diseases;
* Evidence of other clinically significant uncontrolled condition(s) such as uncontrolled and/or active systemic infection (viral, bacterial or fungal)
* A history of other malignant tumors within the past 5 years, excluding localized thyroid cancer and in situ skin cancer;
* Serum total bilirubin >1.5 ULN (upper limit of normal) (excluding leukemia infiltration); ALT or AST or ALP >5 ULN; serum creatinine >1.5 ULN and creatinine clearance rate <40 mL/min; LVEF <50%;
* Known HIV infection;
* Known central nervous system leukemia infiltration;
* Gastrointestinal diseases known to affect venetoclax absorption as judged by the investigator;
* Inability to understand or comply with the study protocol.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
1-year EFS | 1 year
  1-year event free survival rate

SECONDARY OUTCOMES:
CR/CRi | At the end of Cycle 1 (up to 42 days)
  Complete remission/complete remission with incomplete count recovery
OS | through study completion, up to 3 years
  Overall survival
MRD | At the end of Cycle 1 (up to 42 days)
  Percentage of participants who converted to MRD < 10^-3 after the first cycle of treatment.
Safety of induction therapy | At the end of Cycle 1 (up to 42 days)
  Adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China